CLINICAL TRIAL: NCT05172856
Title: A Phase Ib, Open-Label, Multi-Center, Study of Primary Efficacy and Safety of IBI321 Monotherapy or Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: A Phase Ib Study of Primary Efficacy and Safety of IBI321 Monotherapy or Combination Therapy in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI321A103
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI321 in advanced solid tumors (Experimental)
  Interventions: Drug: IBI321

INTERVENTIONS:
Drug: IBI321 — IBI321 at a dose no higher than RP2D, D1 IV Q3W.

SUMMARY:
This is open-label, multicenter, Phase Ib study is designed to evaluate the Primary Efficacy and Safety of IBI321 Monotherapy or Combination Therapy in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Male or female subjects ≥18 years and ≤75 years.
3. At least one measurable lesion per RECIST version 1.1
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
5. Life expectancy of ≥ 12 weeks.
6. Adequate hematologic and end organ function

Exclusion Criteria:

1. Failure to recover from adverse events from the most recent anti-tumor treatments
2. Acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
3. Subjects with CNS metastasis unless they are asymptomatic or adequately treated with radiotherapy and/or surgery and subjects are neurologically stable with minimal residual symptoms/signs.
4. Any other serious underlying medical (e.g., uncontrolled hypertension, active uncontrolled infection, active gastric ulcer,uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, other serious cardiac conditions not listed in exclusion criteria), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.
5. Pregnancy, lactation, breastfeeding.
6. Previous exposure to any anti-TIGIT antibody, or recombinant protein.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators. | From Baseline until disease progression (up to 2 years)

SECONDARY OUTCOMES:
Progression Free Survival (PFS), According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators. | From Baseline until disease progression (up to 2 years)
Overall Survival (OS) | From Day 1 to up to 2 years
Percentage of Participants with Adverse Events (AEs) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 | From Day 1 to up to 2 years
Area Under the Concentration-Time Curve (AUC) of IBI321 | From Day 1 up to 2 years
Maximum Serum Concentration (Cmax) of IBI321 | From Day 1 up to 2 years
Minimum Serum Concentration (Cmin) of IBI321 | From Day 1 up to 2 years
Clearance (CL) of IBI321 | From Day 1 up to 2 years
Percentage of Participants with Anti-Drug Antibodies (ADAs) to IBI321 | From Day 1 up to 2 years
Percentage of Participants with Neutralizing Antibody (Nab) to IBI321 | From Day 1 up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No